CLINICAL TRIAL: NCT04951219
Title: A 52-Week, Phase 3, Open-Label Extension Study, With a Double-blind Lead-in, to Evaluate Safety and Biomarkers of Resmetirom (MGL-3196) in Patients With Non-alcoholic Fatty Liver Disease (NAFLD), MAESTRO-NAFLD-Open-Label-Extension (MAESTRO-NAFLD-OLE)
Brief Title: A Phase 3 Study to Evaluate Safety and Biomarkers of Resmetirom (MGL-3196) in Patients With Non-alcoholic Fatty Liver Disease (NAFLD), MAESTRO-NAFLD-Open-Label-Extension (MAESTRO-NAFLD-OLE)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Madrigal Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MGL-3196-18
Record Dates: First submitted 2021-06-18; First posted 2021-07-06 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD; NASH; Hyperlipidemia; Resmetirom; Thyroid hormone receptor beta; Hepatic; Fibrosis; NASH resolution; Thyroid hormone receptor agonist; Cardiovascular; Dyslipidemia; Fatty liver disease; Nonalcoholic steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hyperlipidemias; Thyroid Hormone Resistance Syndrome; Fibrosis; Dyslipidemias | interventions — resmetirom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Select patients will be randomized in 1:1 manner to a double-blind, 12-week lead-in treatment period. Only investigators, patients, and the Sponsor will be blinded to treatment assignment during the double-blind treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Double-blind 80 mg Daily (Experimental): For patients assigned to double-blind treatment and who completed Week 52 and 56 of MAESTRO-NAFLD-1, double-blind resmetirom 80 mg for first 12 weeks followed by open-label resmetirom 100 mg for weeks 12-52
  Interventions: Drug: Resmetirom
- Double-blind 100 mg Daily (Experimental): For patients assigned to double-blind treatment and who completed Week 52 and 56 of MAESTRO-NAFLD-1, double-blind resmetirom 100 mg for first 12 weeks followed by open-label resmetirom 100 mg for weeks 12-52
  Interventions: Drug: Resmetirom
- Open-label (Experimental): For patients assigned to open-label treatment and who completed Week 52 and 56 of MAESTRO-NAFLD-1, open-label resmetirom at same dose as MGL-3196-14 for an additional 52 weeks. NASH cirrhosis patients may receive open-label resmetirom for an additional 52 weeks (ie, 52 weeks in MGL-3196-14 and 104 weeks in MGL-3196-18).
  Interventions: Drug: Resmetirom
- Open-Label 80 mg (Experimental): For patients with NASH cirrhosis who were screen failures from MGL-3196-11, open-label resmetirom 80 mg for 104 weeks
  Interventions: Drug: Resmetirom
- Open Label 100 mg (Experimental): For patients without NASH cirrhosis who were screen failures from MGL-3196-11, open-label resmetirom 100 mg for 52 weeks
  Interventions: Drug: Resmetirom
- Open-Label 40 mg (Experimental): For NASH cirrhosis patients who enter MGL-3196-18 directly or were screen failures from MGL-3196-19, open-label resmetirom 40 mg for 104 weeks
  Interventions: Drug: Resmetirom

INTERVENTIONS:
Drug: Resmetirom — Tablet
  Other Names: MGL-3196

SUMMARY:
A 52-Week, Multi-center, Open-label, Active Treatment Extension Study to Evaluate Safety and Tolerability of Once Daily, Oral Administration of Resmetirom (MGL-3196)

ELIGIBILITY:
Inclusion Criteria:

* For patients who completed MAESTRO-NAFLD-1, completed the Week 52 visit, and completed the Week 56 visit within 90 days of the Extension Day 1 visit, and are willing to participate in MAESTRO-NAFLD-OLE and provide written informed consent.
* For patients who screen failed MAESTRO-NASH, must provide written informed consent for MAESTRO-NAFLD-OLE and must have screened and met all eligibility requirements for MAESTRO-NASH within 90 days of the Extension Day 1 visit for MAESTRO-NAFLD-OLE and have a liver biopsy that is ineligible for MAESTRO-NASH within 6 months of the Extension Day 1 visit. Eligible liver biopsy for MAESTRO-NAFLD-OLE must have one of the following results:

  * NAS = 3, steatosis 1, ballooning 1, inflammation 1, OR NAS = 3, ballooning 0, with F1B, F2 or F3
  * NAS ≥ 4, at least 1 in all NAS components, F1A or F1C, PRO-C3 ≤ 14 (NASH, but ineligible for MAESTRO-NASH)
  * Compensated NASH cirrhosis based on biopsy at screening of MAESTRO-NASH and baseline of MAESTRO-NAFLD-OLE, including Child Pugh-A (score 5-6), MELD <12, albumin ≥3.2, and bilirubin <2
* For patients who screen failed from MAESTRO-NASH OUTCOMES and de novo patients, must have documented CP-A/B (score <8) NASH cirrhosis (including minimal decompensation) and MELD <15 unless MELD >=15 based on non-cirrhotic parameters. MAESTRO-NASH OUTCOMES screen failures must have screened and met all eligibility requirements for MAESTRO-NASH OUTCOMES within 90 days of the Extension Day 1 visit for MAESTRO-NAFLD-OLE .

Exclusion Criteria:

* A history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to Extension Day 1.
* Diagnosis of hepatocellular carcinoma or other carcinomas that may prevent participation in the Extension study.
* Chronic liver diseases
* Has an active autoimmune disease
* Any other condition which, in the opinion of the Investigator, would impede compliance, hinder completion of the study, compromise the well-being of the patient, or interfere with the study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The effect of once daily, oral administration of resmetirom on the incidence of adverse events. | 52 weeks

SECONDARY OUTCOMES:
Percent change in the hepatic fat fraction as determined by MRI-PDFF from baseline | 16 weeks
Percent change in the hepatic fat fraction as determined by MRI-PDFF from baseline | 52 weeks
Percent change in LDL-C from baseline | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Taub, MD, Study Director — Madrigal Pharmaceuticals, Inc.
Locations (71):
- United States (70):
  - Central Research Associates, Birmingham, Alabama
  - Arizona Liver Health - Chandler, Chandler, Arizona
  - East Valley Family Physicians, Chandler, Arizona
  - The Institute For Liver Health - Glendale, Glendale, Arizona
  - The Institute For Liver Health - Tucson, Tucson, Arizona
  - Adobe Gastroenterology, Tucson, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Fresno Clinical Research Center, Fresno, California
  - National Research Institute - Huntington Park, Huntington Park, California
  - Ruane Clinical Research Group, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - National Research Institute - Los Angeles, Los Angeles, California
  - National Research Institute - Panorama City, Panorama City, California
  - San Fernando Valley Health Institute, West Hills, California
  - South Denver Gastroenterology - Swedish Medical Center Office, Englewood, Colorado
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Covenant Research, Fort Myers, Florida
  - Velocity Clinical Research, Hallandale Beach (MD Clinical), Hallandale, Florida
  - Floridian Clinical Research, Hialeah, Florida
  - Nature Coast Clinical Research - Inverness, Inverness, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Orlando Research Center, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Covenant Research, Sarasota, Florida
  - The Villages Research Center, The Villages, Florida
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Chicago Research Center, Chicago, Illinois
  - Northwestern Memorial Physicians Group, Chicago, Illinois
  - Iowa Diabetes Research, West Des Moines, Iowa
  - Kansas Medical Clinic - Gastroenterology, Topeka, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Digestive Health Center of Louisiana, Baton Rouge, Louisiana
  - Tandem Clinical Research - New Orleans Area Site, Marrero, Louisiana
  - Clinical Trials of America, West Monroe, Louisiana
  - Gastrointestinal Associates & Endoscopy Center - Flowood, Flowood, Mississippi
  - Southern Therapy and Advanced Research, Jackson, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Henderson Research Center, Henderson, Nevada
  - Clarity Clinical Research, East Syracuse, New York
  - Mount Sinai Health System, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cumberland Research Associates, Fayetteville, North Carolina
  - Diabetes and Endocrinology Consultants, Morehead City, North Carolina
  - Aventiv Research Columbus, Columbus, Ohio
  - Awasty Research Network, Marion, Ohio
  - Premier Medical Group - Clarksville - Dunlop Lane, Clarksville, Tennessee
  - Gastro One - Germantown Office - Wolf Park Drive, Germantown, Tennessee
  - Pinnacle Clinical Research - Austin, Austin, Texas
  - The Liver Institute At Methodist Dallas, Dallas, Texas
  - Dallas Research Center, Dallas, Texas
  - Liver Center of Texas, Dallas, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Texas Digestive Disease Consultants, Fort Worth, Texas
  - Liver Associates of Texas, Houston, Texas
  - Doctor's Hospital at Renaissance, McAllen, Texas
  - Plano Research Center, Plano, Texas
  - Texas Liver Institute/American Research Corporation, San Antonio, Texas
  - Pinnacle Clinical Research - San Antonio, San Antonio, Texas
  - San Antonio Research Center, San Antonio, Texas
  - Texas Digestive Disease Consultants - San Marcos, San Marcos, Texas
  - Impact Research Institute, Waco, Texas
  - Texas Digestive Disease Consultants - Bay Area Houston Endoscopy Center, Webster, Texas
  - Wasatch Peak Family Practice, Layton, Utah
  - Salt Lake City Research Center, Murray, Utah
  - Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - National Clinical Research - Richmond, Richmond, Virginia
  - Virginia Commonwealth University School of Medicine, Richmond, Virginia
  - Liver Institute Northwest, Seattle, Washington
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico

REFERENCES:
- [Derived] Harrison SA, Ratziu V, Anstee QM, Noureddin M, Sanyal AJ, Schattenberg JM, Bedossa P, Bashir MR, Schneider D, Taub R, Bansal M, Kowdley KV, Younossi ZM, Loomba R. Design of the phase 3 MAESTRO clinical program to evaluate resmetirom for the treatment of nonalcoholic steatohepatitis. Aliment Pharmacol Ther. 2024 Jan;59(1):51-63. doi: 10.1111/apt.17734. Epub 2023 Oct 2. PMID 37786277